CLINICAL TRIAL: NCT01942473
Title: Effects of Automated Adjustment of Inspired Oxygen on Fluctuations of Regional Cerebral and Arterial Oxygenation in Preterm Infants With Frequent Desaturations
Brief Title: Effects of Automated Adjustment of FiO2 on Cerebral and Arterial Oxygenation in Preterm Infants
Acronym: FiO2-Contr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Helmut Hummler, Chief Division of Neonatology and Pediatric Critical Care, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FiO2_Ulm
Record Dates: First submitted 2012-08-03; First posted 2013-09-16 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Preterm Infant; RDS
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automated FiO2 control (Experimental): Infants will be changed to a specific ventilator device approved for clinical use in neonates in Germany (Avea, Carefusion 234 GmbH Hoechberg, Germany), which is capable to automatically adjust the FiO2 based on readings of an incorporated SpO2 monitoring device. Infants will be allowed to adjust for at least 2h using the ventilator settings as chosen by the clinical team responsible. Thereafter, data will be recorded for 24h experimental time.
  Interventions: Device: Automated FiO2 Control
- Manual Adjustment (Placebo Comparator): Infants will be exposed to the first study phase (clinical routine or automated FiO2 adjustment) for 24 h and then will be switched to the alternate mode (automated FiO2 adjustment or clinical routine) for another 24 h.

INTERVENTIONS:
Device: Automated FiO2 Control — Infants will be ventilated with or without automated FiO2-Control in a randomized sequence.
  Arms: Automated FiO2 control

SUMMARY:
In this study the investigators test the hypothesis that automated FiO2 adjustment increases the time of brain tissue oxygenation within the intended reference range. Furthermore, the investigators studied the change in workload during automated FiO2 adjustment as compared to manual adjustment by the nursing staff.

DETAILED DESCRIPTION:
Recorded data on brain tissue oxygenation will be compared with reference data obtained from other studies. Data from experimental mode (automated FiO2 control will be compared with manual FiO2 control).

ELIGIBILITY:
Inclusion Criteria:

* postmenstrual age <30 wks GA at study time
* on nasal/nasopharyngeal CPAP or mechanical ventilation (including nasopharyngeal IMV)
* at least 4 desaturations (SpO2 <80%) during an 8 hour period within the 24h before the study using a standard pulse oximeter incorporated in the NICU (Dash 3000, General Electric, Freiburg; 10s averaging time, delay 10s)

Exclusion Criteria:

* postnatal age <96h (to exclude rapidly changing conditions during the early phase of RDS and to avoid handling of the infant during the critical period for IVH)
* congenital cyanotic heart disease
* no decision for full treatment support
* Average FiO2 during the last 24h bevor the active study phase >0.60
* Congenital malformations of the lung or the diaphragm (i.e. diaphragmatic hernia, congentital cystic lung diseases...)
* Clinically clear evidence for seizures
* Ongoing Sepsis (CRP > 10mg/l, or positive blood culture, requirement of catecholamines)
* Need of blood-transfusion during study

Ages: 96 Hours to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation | 48 hours
  mean cerebral tissue oxygen saturation as well als distribution of cerebral tissue oxygen saturation over time will be assessed

SECONDARY OUTCOMES:
number and mean duration of episodes with an SpO2 <80%, <75%, <70% and with hyperoxemia (SpO2 >96%) | 48 hours
  The number and mean duration of expisodes of desaturation and with hyperoxemia will be assessed
time within a defined target range of cerebral oxygen saturation (59% - 81%) | 48 hours
  time (as measured as the percentage of the total recording time) within a defined target range of cerebral oxygen saturation (59% - 81%) which corresponds to the 10th and 90th percentile obtained from a pilot study in 16 preterm infants with desaturations during the time when their SpO2 was aimed within the target range of a SpO2 of (88-96%).
workload for the medical staff related to number of adjustments of FiO2 | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Markus Waitz, MD, Principal Investigator — Children's Hospital, University of Ulm
Locations (1):
- Children's Hospital University of Ulm, Ulm, Germany

REFERENCES:
- [Derived] Waitz M, Schmid MB, Fuchs H, Mendler MR, Dreyhaupt J, Hummler HD. Effects of automated adjustment of the inspired oxygen on fluctuations of arterial and regional cerebral tissue oxygenation in preterm infants with frequent desaturations. J Pediatr. 2015 Feb;166(2):240-4.e1. doi: 10.1016/j.jpeds.2014.10.007. Epub 2014 Nov 18. PMID 25454938